CLINICAL TRIAL: NCT00221936
Title: Patient Controlled Oral Analgesia (PCOA) for Postoperative Pain Management After Total Knee Replacement-A Pilot Study
Brief Title: Patient Controlled Oral Analgesia for Postoperative Pain Management After Total Knee Replacement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Patti Kastanias, University Health Network
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UHN04-0394-AE
Record Dates: First submitted 2005-09-20; First posted 2005-09-22 (Estimated); Last update posted 2008-12-05 (Estimated); Status verified 2005-07

CONDITIONS: Self-Administered Versus Nurse Administered Pain Medication.
MeSH Terms: interventions — Self Administration

INTERVENTIONS:
Behavioral: Self-administration or nurse administered medication

SUMMARY:
Patient Centered Care (PCC) is "an approach that consciously adopts the patient's perspective...about what matters" (Gerteis, Edgeman, Levitan, Walker, Stokes, Cleary, Delbanco, 1993). Experiencing pain is the most common concern of patients before surgery - even ahead of whether the surgery would improve their condition (Apfelbaum, 2003). Current standard of practice for post-operative pain management in most acute care hospitals today is intravenous patient controlled analgesia (IV PCA). However, despite the fact that patients prefer IV PCA because it affords them greater control and provides them with better pain relief (Ballantyne, Carr, deFerranti, Suarez, Lau, Chalmers, Angelillo, Mosteller, 1998 ; Rawal, 2001), hospitals routinely take control of pain medications away from patients once they are switched to pain tablets. Patients must then wait, in pain, for their nurse to bring them pain tablets.

Patient controlled oral analgesia (PCOA) has been utilitzed in several centers in the US and Germany. Preliminary evidence from the literature seems to indicate that the benefits of PCOA are similar to IV PCA including increased patient satisfaction and better pain control (Striebel, Romer, Kopf, Schwagmeier ,1996; Striebel, Scheitza, Philippi, Behrens, Toussaint, 1998). At the Toronto Western Hospital, University Health Network, we have successfully implemented a PCOA program on two surgical units (Orthopedics/Rheumatology and Spinal). The purpose of this study is to compare usual nurse administered oral analgesia to PCOA with respect to pain, patient satisfaction, and passive range of knee motion in postoperative total knee replacement patients.

ELIGIBILITY:
Inclusion Criteria:

* able to read and write English
* post elective total knee replacement surgery (primary or revision)
* already on IV PCA
* age 18-80
* able to tolerate oral medication
* able to physically open a childproof vial independently (including the absence of any significant problems with manual power, dexterity or visual acuity)
* able and willing to complete Oral PCA flowsheet

Exclusion Criteria:

* history of substance abuse
* history of sleep apnea
* episode(s) of confusion, disorientation during this admission
* episode(s) of respiratory depression during this admission
* history of major psychiatric disorder pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2004-07; Primary Completion 2005-07 (Actual); Study Completion 2005-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patti Kastanias, RN, MSc(A), ACNP, Principal Investigator — University of Health Network, Toronto
Locations (3):
- Canada (3):
  - Toronto Western Hospital, Toronto, Ontario
  - University Health Network, Toronto, Ontario
  - Universtiy Health Network, Toronto, Ontario